CLINICAL TRIAL: NCT01078246
Title: Post-Licensure Safety Study of ISENTRESS™ in a US Managed Care Network
Brief Title: Post-Licensure Safety Study of ISENTRESS™ (Raltegravir) in a United States Managed Care Network (MK-0518-268)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 0518-268; EP08025.006 (Other: Merck); 2010_021 (Other: Merck)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: HIV-1 Infections
Keywords: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- Raltegravir Cohort Only: Participants with HIV-1 infection who received raltegravir (RAL) on or after 12 October 2007 (the market authorization date in the United States) (Raltegravir Cohort). These participants contributed data to the Raltegravir Cohort only.
- Historical and Raltegravir Cohorts Only: Participants with HIV-1 infection who 1) received antiretroviral therapy (non-RAL) between 1 January 2005 and 11 October 2007 (Historical Cohort), and 2) received RAL on or after 12 October 2007 (Raltegravir Cohort). These participants contributed data to the Historical and Raltegravir Cohorts only.
- Historical Cohort Only: Participants with HIV-1 infection who received antiretroviral therapy (non-RAL) between 1 January 2005 and 11 October 2007 (Historical Cohort). These participants contributed data to the Historical Cohort only.
- Historical and Concurrent Cohorts Only: Participants with HIV-1 infection who 1) received antiretroviral therapy (non-RAL) between 1 January 2005 and 11 October 2007 (Historical Cohort), and 2) received therapy with a new non-RAL antiretroviral therapy after 12 October 2007 (Concurrent Cohort). These participants contributed data to the Historical and Concurrent Cohorts only.
- Concurrent Cohort Only: Participants with HIV-1 infection who received therapy with a new non-RAL antiretroviral therapy after 12 October 2007 (Concurrent Cohort). These participants contributed data to the Concurrent Cohort only.
- Concurrent and Raltegravir Cohorts Only: Participants with HIV-1 infection who 1) received therapy with a new non-RAL antiretroviral therapy on or after 12 October 2007 (Concurrent Cohort), and 2) received RAL after 12 October 2007 (Raltegravir Cohort). These participants contributed data to the Concurrent and Raltegravir Cohorts only.
- Historical, Concurrent and Raltegravir Cohorts: Participants with HIV-1 infection who 1) received antiretroviral therapy (non-RAL) between 1 January 2005 and 11 October 2007 (Historical Cohort), 2) received therapy with a new non-RAL antiretroviral therapy on or after 12 October 2007 (Concurrent Cohort), and 3) received RAL after 12 October 2007 (Raltegravir Cohort). These participants contributed data to all three cohorts.

SUMMARY:
The objective of this study is to monitor Health Outcomes of Interest (HOI) in participants with human immunodeficiency virus-1 (HIV-1) infection following treatment with Raltegravir.

DETAILED DESCRIPTION:
Study participants contributed data to one or more of 3 cohorts: 1) Historical Cohort: HIV-infected participants treated with antiretroviral therapy in the course of ordinary clinical practice at the clinics and medical centers of Kaiser Permanente (KP) between 1 January 2000 and 12 October 2007 (date of market authorization for raltegravir in USA), 2) Concurrent Cohort: HIV-infected participant treated with a new non-raltegravir antiretroviral therapy in the course of ordinary clinical practice at the clinics and medical centers of KP on or after 12 October 2007, and 3) Raltegravir Cohort: HIV-infected participant treated with raltegravir in the course of ordinary clinical practice at the clinics and medical centers of KP on or after 12 October 2007. Participants could contribute data to more than one cohort, but no overlap in follow-up time was allowed.

ELIGIBILITY:
Inclusion Criteria:

* Historical Cohort: HIV-infected participant treated with antiretroviral therapy in the course of ordinary clinical practice at the clinics and medical centers of Kaiser Permanente (KP) between 1 January 2000 and 12 October 2007 (date of market authorization for raltegravir in USA)
* Raltegravir Cohort: HIV-infected participant treated with raltegravir in the course of ordinary clinical practice at the clinics and medical centers of KP on or after 12 October 2007
* Concurrent Cohort: HIV-infected participant treated with a new non-raltegravir antiretroviral therapy in the course of ordinary clinical practice at the clinics and medical centers of KP on or after 12 October 2007
* All participants must have at least one year of continuous membership with KP prior to date when the participant received the first dispensed prescription for study drug (index date) to allow for the assessment of medical and treatment history

Exclusion Criteria:

* Less than 18 years of age
* Do not receive their medications through the KP pharmacy system
* Do not receive their laboratory examinations through the KP system
* Participating in the raltegravir phase III or expanded access program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years old and older
Sampling Method: Non-Probability Sample
Enrollment: 7124 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2014-12-09 (Actual); Study Completion 2014-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: EUPAS Register (EUPAS17981) — http://www.encepp.eu/encepp/viewResource.htm?id=17982

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The analyses in this study are based on data collected from a cohort of human immunodeficiency virus (HIV-1)-infected participants in a setting of routine clinical care at the Kaiser Permanente medical centers in California, United States. Participants could contribute data to more than one cohort, but no overlap in follow-up time was allowed.
Period: Overall Study
Arm/Group | Raltegravir Cohort Only | Historical and Raltegravir Cohorts Only | Historical Cohort Only | Historical and Concurrent Cohorts Only | Concurrent Cohort Only | Concurrent and Raltegravir Cohorts Only | Historical, Concurrent and Raltegravir Cohorts
Started | 1041 | 405 | 1963 | 152 | 3310 | 231 | 22
Completed | 1041 | 405 | 1963 | 152 | 3310 | 231 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Cohort Only | Historical and Raltegravir Cohorts Only | Historical Cohort Only | Historical and Concurrent Cohorts Only | Concurrent Cohort Only | Concurrent and Raltegravir Cohorts Only | Historical, Concurrent and Raltegravir Cohorts | Total
Number analyzed (Participants) | 1041 | 405 | 1963 | 152 | 3310 | 231 | 22 | 7124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (10.7) | 49.2 (10.0) | 45.8 (10.1) | 44.9 (9.9) | 43.0 (11.5) | 46.8 (12.4) | 45.5 (9.9) | 45.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 41 | 195 | 23 | 340 | 33 | 4 | 757
  Male | 920 | 364 | 1768 | 129 | 2970 | 198 | 18 | 6367

OUTCOME MEASURES:

1. Primary Outcome: Incidence of AIDS-defining and Non-AIDS-defining Malignancy
Description: All new malignancies occurring during the risk period, including Acquired Immune Deficiency Syndrome (AIDS)-defining and non-AIDS-defining malignancies, were identified through the Kaiser Permanente cancer registries. The registry data was supplemented by the use of computer-stored records of outpatient visits, Emergency Department visits and hospitalizations to identify cancers that would not be captured through the cancer registries (e.g. cutaneous Kaposi's sarcoma).The AIDS-defining malignancies reported for any cohort were invasive cervical cancer, Kaposi's sarcoma, and non-Hodgkin lymphoma. Incidence is reported as unadjusted, crude rates.
Time Frame: Historical Cohort: up to 33 months (January 2005 to October 2007); Raltegravir and Concurrent Cohorts: up to 69 months (October 2007 to June 2013)
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Groups:
- Raltegravir Cohort: Participants with HIV-1 infection who received RAL on or after 12 October 2007. Participants from the Historical Cohort and the Concurrent Cohort were eligible for inclusion in the Raltegravir Cohort.
- Historical Cohort: Participants with HIV-1 infection who received antiretroviral therapy (non-RAL) between 1 January 2005 and 11 October 2007. These participants were eligible for inclusion in the Concurrent and Raltegravir Cohorts.
- Concurrent Cohort: Participants with HIV-1 infection who received therapy with a new non-RAL antiretroviral therapy after 12 October 2007. Participants from the Historical Cohort were eligible for inclusion in the Concurrent Cohort. Participants from the Concurrent Cohort were eligible for inclusion in the Raltegravir Cohort.
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup
  AIDS-defining Malignancy | 13.0 [9.6 to 16.3] | 8.9 [5.7 to 12.2] | 9.3 [7.4 to 11.2]
  Non-AIDS-defining Malignancy | 18.2 [14.3 to 22.1] | 9.1 [5.8 to 12.3] | 10.3 [8.3 to 12.3]
Statistical Analysis 1: Comparison: Raltegravir Cohort vs Historical Cohort; AIDS-defining malignancies; Test type: Superiority or Other; p = 0.002, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 2.282, 95% CI 2-sided [1.344 to 3.875]
Statistical Analysis 2: Comparison: Raltegravir Cohort vs Historical Cohort; AIDS-defining malignancies; Test type: Superiority or Other; p < 0.05, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 2.840, 95% CI 2-sided [1.621 to 4.977]
Statistical Analysis 3: Comparison: Raltegravir Cohort vs Concurrent Cohort; AIDS-defining malignancies; Test type: Superiority or Other; p = 0.005, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.871, 95% CI 2-sided [1.207 to 2.899]
Statistical Analysis 4: Comparison: Raltegravir Cohort vs Concurrent Cohort; AIDS-defining malignancies; Test type: Superiority or Other; p = 0.004, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.879, 95% CI 2-sided [1.227 to 2.879]
Statistical Analysis 5: Comparison: Raltegravir Cohort vs Historical Cohort; Non-AIDS-defining malignancies; Test type: Superiority or Other; p = 0.008, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.943, 95% CI 2-sided [1.191 to 3.168]
Statistical Analysis 6: Comparison: Raltegravir Cohort vs Historical Cohort; Non-AIDS-defining malignancies; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 2.459, 95% CI 2-sided [1.454 to 4.159]
Statistical Analysis 7: Comparison: Raltegravir Cohort vs Concurrent Cohort; Non-AIDS-defining malignancies; Test type: Superiority or Other; p = 0.004, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.776, 95% CI 2-sided [1.199 to 2.631]
Statistical Analysis 8: Comparison: Raltegravir Cohort vs Concurrent Cohort; Non-AIDS-defining malignancies; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.860, 95% CI 2-sided [1.274 to 2.717]

2. Primary Outcome: Incidence of Clinically Important Hepatic Events
Description: Hepatic events occurring during the risk period were identified through computer-stored records of laboratory values, outpatient visits, Emergency Department visits, and hospitalizations. Significant hepatic events were identified based on algorithms utilizing a combination of diagnoses, procedures, and laboratory results. Incidence is reported as unadjusted, crude rates.
Time Frame: as for outcome 1
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup | 19.0 [14.9 to 23.0] | 25.0 [19.6 to 30.5] | 17.1 [14.5 to 19.7]
Statistical Analysis 1: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.255, Poisson regression; The analysis included adjustments for raltegravir exposure, propensity score, treatment regimen (1st, 2nd, 3rd+), and Hepatitis B/C status; Incidence Rate Ratio = 0.807, 95% CI 2-sided [0.557 to 1.168]
Statistical Analysis 2: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.646, Cox Proportional Hazard Regression; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.907, 95% CI 2-sided [0.597 to 1.376]
Statistical Analysis 3: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.182, Poisson Regression; [statistical method as in outcome 2, analysis 1]; Incidence Rate Ratio = 1.268, 95% CI 2-sided [0.895 to 1.795]
Statistical Analysis 4: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.188, Cox Proportional Hazard Regression; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.257, 95% CI 2-sided [0.894 to 1.768]

3. Primary Outcome: Incidence of Clinically Important Skin Events
Description: Significant skin events (e.g. Stevens-Johnson syndrome and toxic epidermal necrolysis) occurring during the risk period were identified through the use of computer-stored records of outpatient visits, Emergency Department visits and hospitalizations. The identification of potential significant skin events was based on algorithms utilizing a combination of diagnoses, procedures and/or medications. Surveillance of outpatient visits was limited to rashes coded as drug-related and requiring use of steroid (e.g. prednisone) administration. Incidence is reported as unadjusted, crude rates.
Time Frame: as for outcome 1
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup | 40.6 [34.4 to 46.8] | 69.8 [60.4 to 79.2] | 63.6 [58.2 to 69.1]
Statistical Analysis 1: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.897, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.016, 95% CI 2-sided [0.796 to 1.297]
Statistical Analysis 2: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.070, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.287, 95% CI 2-sided [0.980 to 1.690]
Statistical Analysis 3: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.575, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.067, 95% CI 2-sided [0.850 to 1.339]
Statistical Analysis 4: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.626, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.057, 95% CI 2-sided [0.847 to 1.319]

4. Primary Outcome: Incidence of Clinically Important Muscle Events
Description: Significant muscle events (e.g. rhabdomyolysis) occurring during the risk period were identified through the use of computer-stored records of laboratory values, outpatient visits, Emergency Department visits and hospitalizations. The identification of potential significant muscle events was based on algorithms utilizing a combination of diagnoses, procedures and/or laboratory results for creatinine kinase. The number of muscle events did not meet the threshold for statistical analysis per protocol. Incidence is reported as unadjusted, crude rates.
Time Frame: as for outcome 1
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup | 3.4 [1.7 to 5.1] | 3.3 [1.4 to 5.3] | 1.5 [0.7 to 2.3]

5. Primary Outcome: Incidence of Lipodystrophy
Description: Lipodystrophy (e.g. lipoatrophy, facial wasting) occurring during the risk period was identified through the use of computer-stored records of outpatient visits, Emergency Department visits and hospitalizations. The identification of potential lipodystrophy was based on two coded diagnoses codes indicative of lipodystrophy appearing at least 6 months apart over the course of patient care, the identification of interventions to treat such conditions (e.g. sculptra therapy), or procedural codes for Computerized Tomography indicating incident neck or abdominal lipoaccumulation. Incidence is reported as unadjusted, crude rates.
Time Frame: as for outcome 1
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup | 20.6 [15.9 to 25.4] | 35.6 [28.9 to 42.4] | 9.2 [7.2 to 11.1]
Statistical Analysis 1: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p < 0.0001, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 0.389, 95% CI 2-sided [0.274 to 0.551]
Statistical Analysis 2: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p < 0.05, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 0.471, 95% CI 2-sided [0.314 to 0.707]
Statistical Analysis 3: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.015, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.650, 95% CI 2-sided [1.102 to 2.470]
Statistical Analysis 4: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.018, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.622, 95% CI 2-sided [1.085 to 2.425]

6. Secondary Outcome: Incidence of Clinically Important Cardiovascular Events
Description: Significant cardiovascular events occurring during the risk period were identified through the use of computer-stored records and defined as inpatient events based on algorithms that utilize a combination of diagnosis and/or procedure codes. The identification of potential significant cardiovascular events was based on the occurrence of major adverse cardiovascular events (MACE) which include acute myocardial infarction (MI), ischemic stroke, unstable angina, revascularization (e.g. percutaneous coronary intervention (PCI) and coronary bypass graft surgery (CABG)), and cardiovascular death. Incidence is reported as unadjusted, crude rates.
Time Frame: as for outcome 1
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup | 6.7 [4.4 to 9.1] | 6.4 [3.7 to 9.1] | 4.0 [2.8 to 5.3]
Statistical Analysis 1: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.423, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 0.750, 95% CI 2-sided [0.370 to 1.517]
Statistical Analysis 2: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.631, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.208, 95% CI 2-sided [0.559 to 2.612]
Statistical Analysis 3: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.592, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 0.845, 95% CI 2-sided [0.458 to 1.561]
Statistical Analysis 4: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.943, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.022, 95% CI 2-sided [0.565 to 1.850]

7. Secondary Outcome: Incidence of All-cause Mortality
Description: All-cause mortality occurring during the risk period was identified through the use of computer-stored records of Emergency Department visits, hospitalizations, and state death certificates. Deaths were identified from administrative Kaiser Permanente databases, including Kaiser Permanente regional research and respective state(s) mortality files as well as the Social Security Administrative files. Incidence is reported as unadjusted, crude rates.
Time Frame: as for outcome 1
Population: The analysis includes all eligible participants.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person-years of followup
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1699 | 2542 | 3715
Events per 1000 person-years of followup | 16.9 [13.3 to 20.6] | 18.4 [13.7 to 23.0] | 7.7 [6.0 to 9.4]
Statistical Analysis 1: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.109, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 0.708, 95% CI 2-sided [0.464 to 1.080]
Statistical Analysis 2: Comparison: Raltegravir Cohort vs Historical Cohort; Test type: Superiority or Other; p = 0.356, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.486 to 1.296]
Statistical Analysis 3: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.039, Poisson Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Incidence Rate Ratio = 1.556, 95% CI 2-sided [1.022 to 2.370]
Statistical Analysis 4: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.033, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, propensity score, and treatment regimen (1st, 2nd, 3rd+); Hazard Ratio (HR) = 1.564, 95% CI 2-sided [1.036 to 2.361]
Statistical Analysis 5: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.125, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, and propensity score, and was stratified by the 1st treatment regimen; Hazard Ratio (HR) = 1.720, 95% CI 2-sided [0.861 to 3.437]
Statistical Analysis 6: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.881, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, and propensity score, and was stratified by the 2nd treatment regimen; Hazard Ratio (HR) = 1.056, 95% CI 2-sided [0.517 to 2.155]
Statistical Analysis 7: Comparison: Raltegravir Cohort vs Concurrent Cohort; Test type: Superiority or Other; p = 0.107, Cox Proportional Hazard Regression; The analysis included adjustments for raltegravir exposure, and propensity score, and was stratified by the 3rd+ treatment regimen; Hazard Ratio (HR) = 2.077, 95% CI 2-sided [0.854 to 5.05]

ADVERSE EVENTS:
Description: Per protocol, adverse events were not collected as part of the study database; therefore, none were collected and the number at risk is zero.
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No